CLINICAL TRIAL: NCT03287180
Title: Adolescent Community Reinforcement Approach (A-CRA) Implementation in Combination With Buprenorphine/Naloxone for Young Adults Ages 18 to 25 With Severe Opioid Use Disorder
Brief Title: Adolescent Community Reinforcement Approach in Combination With Buprenorphine/Naloxone for Severe Opioid Use
Acronym: A-CRA/MAT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to enroll any participants
Sponsor: Emory University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Chestnut Health Systems (Other)
Responsible Party: Principal Investigator, Justine Welsh, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00093907; 1R21DA046738-01 (NIH)
Record Dates: First submitted 2017-09-07; First posted 2017-09-19 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Opioid-Related Disorders; Behavior, Addictive
Keywords: Adolescent Community Reinforcement Approach; A-CRA; Opioid-Related Disorders; Behavior; Psychosocial treatment; Pharmacotherapy; Randomized controlled; Adolescent; Young adult
MeSH Terms: conditions — Opioid-Related Disorders; Behavior, Addictive; Behavior | interventions — Buprenorphine, Naloxone Drug Combination; Naloxone

STUDY DESIGN:
Intervention Model Description: This 12-week randomized controlled pilot trial will begin by an induction on sublingual buprenorphine/naloxone for all participants who would usually receive buprenorphine based treatment in the clinic. After the two-week induction phase, participants will be randomized into two groups. While continuing buprenorphine/naloxone the experimental group will receive a 12-week course of A-CRA, while the control group will be provided medical management by the prescriber. Medical management is the standard treatment approach for prescribing buprenorphine and covers medication adherence, side effects of the medication, assessment of withdrawal/cravings and dose adjustment as indicated. After completion of the 12-week A-CRA intervention, all individuals will receive weekly medical management sessions until week 24 (6 month follow up).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Participants in the experimental group will attend one individual assessment with the study physician for combination of buprenorphine/naloxone 4/1 prescription and urinalysis, along with one weekly Adolescent Community Reinforcement Approach (A-CRA) session (approximately 50 minutes).
  Interventions: Behavioral: Adolescent Community Reinforcement Approach (A-CRA); Other: Combination of buprenorphine/naloxone 4/1
- Control group (Active Comparator): Participants in the control condition will attend weekly individual medical management sessions with the MD who will also provide a prescription for a combination of buprenorphine/naloxone 4/1 (approximately 25 minutes in duration).
  Interventions: Other: Combination of buprenorphine/naloxone 4/1

INTERVENTIONS:
Behavioral: Adolescent Community Reinforcement Approach (A-CRA) — The A-CRA is a modified version of the Community Reinforcement Approach for adolescents and transitional age youth. The A-CRA treatment protocol consists of nineteen procedures designed to promote positive behavior change directed towards prosocial activities and engagement in the individual's community. A community can include but is not limited to: social and peer activities, family interaction, and work or school environments. Some of the highlighted procedures include relapse prevention, sobriety sampling, problem solving, and communication skills. There are also combined parent/and or couples relationship sessions with the young adult. In the current study, 12-weeks of A-CRA treatment will be provided to the intervention group.
  Arms: Experimental group
Other: Combination of buprenorphine/naloxone 4/1 — Buprenorphine is a partial agonist at mu-opioid receptor, an antagonist at kappa-opioid receptor. Naloxone is an antagonist at the mu-opioid receptor. Buprenorphine/naloxone requires the use of an induction to avoid the risk of withdrawal. Participants are instructed not to use opioids for at least 10 hours prior to first dose. Once symptoms of withdrawal score a minimum of 7 on the Clinical Opiate Withdrawal Scale (COWS), the first dose of 4/1 mg will be given. Participants will be monitored for an hour. An additional 4/1 mg dose can be provided to a dose that suppresses withdrawal effects. The physician then provides a prescription for 8/2-16/4 mg for Day 2. Doses can be adjusted with a maximum of total 24/6 mg/day. The target daily dose is 16/4 mg.
  Other Names: Suboxone/Narcan

SUMMARY:
The study assesses whether adding a behavioral intervention, known as the Adolescent Community Reinforcement Approach (A-CRA), to the treatment of individuals already receiving buprenorphine/naloxone can improve treatment success and retention rates in young adults with severe opioid use disorder.

DETAILED DESCRIPTION:
Buprenorphine is one of the medication assisted treatments approved by the FDA for opioid use disorders. Treatment with buprenorphine/naloxone may reduce the risk of opioid overdose and lower the occurrence of further conditions associated with injection drug use such as psychiatric disorders, hepatitis C infection, HIV, and high-risk sexual and criminal behaviors. The study assesses whether adding a behavioral intervention, known as the Adolescent Community Reinforcement Approach (A-CRA), to the treatment of individuals already receiving buprenorphine/naloxone can improve treatment success and retention rates in young adults with severe opioid use disorder.

ELIGIBILITY:
Inclusion Criteria:

* have met DSM-5 criteria for severe opioid use disorder
* no sensitivity to buprenorphine or naloxone
* no further medical/addictive conditions that require immediate medical attention
* ability to read and provide informed consent
* intent to remain in the area for the duration of the study
* able to receive outpatient care
* agreed to use an acceptable birth control method throughout the duration of this study (female participants)

Exclusion Criteria:

* endorsement of imminent and serious suicidality
* medical conditions that take precedence over the presence of treatment for an addictive disorder
* history of an adverse reaction to buprenorphine/naloxone
* current substance use or psychiatric condition requiring a level of care higher than outpatient
* pregnant, nursing or planning pregnancy during the extent of the treatment trial(female participants)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Proportion of opiates-negative urine drug screens over the total number of urine drug screens at each stage | Each session (weekly) up to 24 weeks.
  Qualitative urine test for opiates (+/-) will be performed. All presumptive positive assays will be confirmed by Gas Chromatography-Mass Spectrometry. The concentration value must be greater than or equal to the cutoff to be reported as positive. The opiates test results (positive/negative) will be documented. Proportion of opiates-negative urine drug screens over the total number of urine drug screens at each stage will be reported.
Percent of days of opioid use within the past 90 days as indicated by self-report on the Global Appraisal of Individual Needs | Pre-treatment (baseline) and post-study intervention (12 weeks visit after completion of A-CRA ), and end of follow-up (24-week visit) .
  The Global Appraisal of Individual Needs is a comprehensive, semi-structured interview measure with established validity and reliability used to identify and address a wide range of psychosocial problems in clinical populations. Average administration time for the GAIN Intake version is 1.5 hours and 45 minutes for the follow-up version. The assessment categories include background, school problems, work problems, physical health, sources of stress, risk behaviors and infectious diseases, mental health, substance use, and crime and violence. Substance use categories document self-reported frequency of substance use within the past 90 days for each substance endorsed (alcohol, opioids, marijuana, and other illicit psychoactive drugs). Individuals are able to say that they do not know, or refuse to answer any questions that they do not want to answer.

SECONDARY OUTCOMES:
Completion of the final phase of treatment defined as final study session (yes/no) | 24-week visit
  To investigate any difference in treatment retention in the experimental group compared to the control group.
Number of clinic visits by patient and any expected joint family member sessions | 2-, 12, and 24-week visits.
  To investigate any difference in treatment retention in the experimental group compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Justine Welsh, MD, Principal Investigator — SOM: Psych: Child Psych - CAMP Emory University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Arnett JJ. Emerging adulthood. A theory of development from the late teens through the twenties. Am Psychol. 2000 May;55(5):469-80. PMID 10842426
- [Background] Jones CM, Logan J, Gladden RM, Bohm MK. Vital Signs: Demographic and Substance Use Trends Among Heroin Users - United States, 2002-2013. MMWR Morb Mortal Wkly Rep. 2015 Jul 10;64(26):719-25. PMID 26158353
- [Background] Godley SH, Smith JE, Passetti LL, Subramaniam G. The Adolescent Community Reinforcement Approach (A-CRA) as a model paradigm for the management of adolescents with substance use disorders and co-occurring psychiatric disorders. Subst Abus. 2014;35(4):352-63. doi: 10.1080/08897077.2014.936993. PMID 25035906
- [Background] Wesson DR, Ling W. The Clinical Opiate Withdrawal Scale (COWS). J Psychoactive Drugs. 2003 Apr-Jun;35(2):253-9. doi: 10.1080/02791072.2003.10400007. PMID 12924748
- [Background] Rudd RA, Aleshire N, Zibbell JE, Gladden RM. Increases in Drug and Opioid Overdose Deaths--United States, 2000-2014. MMWR Morb Mortal Wkly Rep. 2016 Jan 1;64(50-51):1378-82. doi: 10.15585/mmwr.mm6450a3. PMID 26720857